CLINICAL TRIAL: NCT03707158
Title: Kids Formats of Anxiety Care Effectiveness Study For Extending the Acceptability and Reach of Services (Kids FACE FEARS)
Brief Title: Kids FACE FEARS Comparative Effectiveness Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Massachusetts General Hospital (Other); South Boston Community Health Center (Other); Johns Hopkins University (Other); Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other); Boston University (Other); Florida International University (Other); University of Washington (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-37862; 6005686 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2018-09-25; First posted 2018-10-16 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Child Anxiety; Anxiety Disorders; Anxiety; Anxiety Symptoms; Anxiety, Mild to Moderate; Pediatric Anxiety Disorders
Keywords: Cognitive Behavioral Therapy (CBT); Online CBT; Telehealth; Anxiety; Child; Therapist-Led CBT; Pediatric Anxiety; Internet-Delivered CBT; iCBT; Telemental Health; Adolescent; Teen; Youth anxiety; Comparative Effectiveness
MeSH Terms: conditions — Anxiety Disorders | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Pragmatic Comparative Effectiveness RCT; Type I Hybrid Effectiveness and Implementation Study
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators (IEs) are masked to treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Online CBT (with minimal therapist involvement) (Active Comparator): The online, multimedia suite of Cool Kids CBT web-based programs for youth anxiety is a supported, self-paced, self-administered online digital CBT anxiety management intervention, with adjunctive therapist phone support. Treatment content runs directly parallel to that included in the therapist-led Cool Kids suite of interventions. Depending on the age of the child, one of two developmentally tailored programs was assigned from the online suite of online Cool Kids interventions (i.e., Cool Kids Online for 7-12 year olds; Chilled Out for 13+ year olds)
  Interventions: Behavioral: Guided Online CBT
- Therapist-Led CBT (telehealth, office-based, or hybrid delivered) (Active Comparator): The Cool Kids suite of therapist-led CBT-based programs for youth anxiety is a well-supported anxiety management intervention, delivered by a therapist across weekly sessions. The therapist-led cognitive-behavioral therapy treatment content runs directly parallel to that included in the Cool Kids online suite of interventions. Depending on the age of the child, one of two developmentally tailored programs was implemented from the suite of therapist-led Cool Kids interventions (i.e., Cool Kids for 7-12 year olds; Chilled for 13-18 year olds). For the present study, Therapist-led CBT could be implemented via telehealth or in-person (i.e., office-based), or as a hybrid format of both telehealth and office-based care. For each therapist-led CBT case, the specific format of care (i.e., telehealth, office-based, or hybrid) was determined via patient/family preferences, collaborative decision-making, hospital policies, and/or COVID-related mandates.
  Interventions: Behavioral: Therapist-Led CBT (telehealth, office-based, or hybrid)

INTERVENTIONS:
Behavioral: Therapist-Led CBT (telehealth, office-based, or hybrid) — Participants receiving therapist-led CBT will participate in therapist-led (telehealth or office-based) CBT treatment for up to 20 weeks. Weekly therapist-led treatment sessions focus on psychoeducation about anxiety, thought challenging and cognitive restructuring, somatic management skills training, youth exposure to feared stimuli, family patterns associated with the maintenance of youth anxiety, and contingent reinforcement.
  Arms: Therapist-Led CBT (telehealth, office-based, or hybrid delivered)
Behavioral: Guided Online CBT — Participants receiving guided online CBT will complete an online, self-paced, standardized and digitalized CBT program for up to 20 weeks with 8 modules, with adjunctive therapist phone support for supportive accountability. The self-administered treatment modules focus on psychoeducation about anxiety, thought challenging and cognitive restructuring, somatic management skills training, youth exposure to feared stimuli, family patterns associated with the maintenance of youth anxiety, and contingent reinforcement.
  Arms: Guided Online CBT (with minimal therapist involvement)

SUMMARY:
The Kids FACE FEARS (Kids Formats of Anxiety Care Effectiveness study For Extending the Acceptability and Reach of Services) is a large-scale, streamlined, pragmatic Randomized Controlled Trial (RCT) evaluating Therapist-Led CBT (telehealth, office-based, or hybrid) vs. Guided Online Cognitive-Behavioral Therapy (CBT) for the treatment of elevated child and adolescent anxiety. Families will be recruited from pediatric health centers serving primarily racial/ethnic minority youth in urban, suburban, and semi-rural regions. Services will be offered in English and Spanish. Patient-centered outcomes will be evaluated across a one-year follow-up period. To compare the effectiveness of the two treatment comparators, investigators will analyze the reports of caregivers, youth, and therapists, as well as independent evaluators who are not informed of each child's treatment assignment. Primary outcomes will focus on family-rated anxiety severity and impairment, treatment responder and remission status rated by independent evaluators, family-perceived effectiveness, and treatment satisfaction. Secondary analyses will examine additional outcomes, predictors of varied outcomes across different subgroups of youth, and facilitators and barriers to treatment implementation. Caregivers, patients, providers, and other key stakeholders will be actively engaged throughout all aspects of the research.

DETAILED DESCRIPTION:
Clinical anxiety is among the most common and impairing psychiatric conditions affecting children and adolescents. Cognitive Behavioral Therapy (CBT) is an effective psychological treatment for youth anxiety, with roughly 60% of youth showing considerable clinical response and global improvements in functioning. Regrettably, despite the existence of well-supported treatments, most youth with anxiety disorders do not receive any form of treatment, especially in resource poor settings.

To extend the reach of CBT, research has provided initial support for several modernized modes of CBT delivery that differentially draw on technology to support varying levels of therapist involvement. For example, telehealth and hybrid options (i.e., mix of telehealth and office-based care) leverage synchronous telecommunications (typically videoconferencing) for the remote provision of live and interactive therapist-led care. Telehealth has been increasingly studied with success as a means to overcome several logistical challenges to traditional brick-and-mortar CBT for youth anxiety and stigma about attending a mental health facility. After years of initial research,m telehealth and hybrid formats became a dominant mode of outpatient mental health care, and in post-pandemic times these formats still play a prominent role (albeit understudied) role in youth mental health care.

Whereas telehealth and hybrid formats offer opportunities to extend the reach of therapist-led CBT, guided online CBT (i.e., self-paced and relatively automated care with minimal therapist involvement) offers a computerized treatment delivery format that reduces therapist demands and person-power needs relative to therapist-led care. For some, guided online CBT may be a more accessible, acceptable, and even effective format, although attrition can be high in self-paced care.

Despite great promise in the use of technology-based strategies for expanding the reach of CBT for pediatric anxiety, much remains to be learned about how such alternative CBT formats perform in typical care settings, what factors may facilitate versus challenge successful implementation and engagement in usual care settings, and whether specific subpopulations of anxious youth may differentially benefit from these options. As with the majority of controlled evidence supporting therapist-led CBT for youth anxiety, most support for telehealth and hybrid CBT has come from trials conducted in tightly controlled contexts and anxiety specialty clinics with highly selected samples and research therapists. Such work cannot speak to the effectiveness of telehealth effectiveness under typical care circumstances. Many of these studies have also been relatively small and underpowered to examine predictors of differential telehealth response. With regard to guided online CBT for pediatric anxiety, research to date has been conducted with predominantly non-Hispanic White and English-speaking samples, and most of the trials have been implemented in anxiety-specialty clinics and/or research settings. Evaluating the effectiveness of guided online CBT in diverse populations under usual care conditions is critical for understanding the extent to which this format can truly expand the accessibility and acceptability of care and reach underserved populations. Furthermore, clinical trials of guided online CBT for anxiety have not included a therapist-led treatment comparison, rendering it hard to make informed comparisons across treatment formats and precluding an understanding of which CBT formats for youth anxiety work best for whom.

The pediatric health care setting offers an optimal public health venue for youth anxiety management, yet there is a critical lack of behavioral health specialty care providers in these settings who are trained in providing mental health treatment, and a lack of information on the optimal methods of treating anxiety in pediatric settings. Accordingly, technology-based treatment options may be a particularly welcome format in pediatric usual care settings..

The Kids FACE FEARS study design entails a large-scale, streamlined, pragmatic, randomized controlled trial (RCT), in which eligible youth with elevated anxiety identified in pediatric health care settings will be randomly assigned to therapist-led CBT (delivered via telehealth, hybrid, or office-based) versus guided online CBT intervention for youth anxiety and monitored for up to one year out. Outcomes for each participant will be monitored across four major assessment points, corresponding to baseline, mid-treatment, post-treatment, and 1 year follow-up. Acute and longer-term outcomes associated with therapist-led versus guided online CBT will be evaluated over a 1-year follow-up period. We will use the well-established Cool Kids suite of therapist-led and online anxiety CBT protocols within pediatric health care networks serving primarily racial-ethnic minority children in both urban and rural settings across four regions of the US: the Northeast, the Mid-Atlantic, the Southeast, and the Pacific Northwest. Natural providers (i.e., not research therapists or anxiety specialists) in these pediatric usual care settings will provide all services. All participants will be identified and referred for enrollment from pediatric health settings. All care and study materials will be provided in English and Spanish.

This study addresses three critical yet unanswered questions related to improving the delivery of modernized CBT formats and treatment outcomes for anxiety in pediatric usual care settings. Answering the following question offers the potential to meaningfully improve the quality of the evidence available to help children, families, and organizational stakeholders make informed, patient-centered decisions regarding clinical practice and implementation strategies for the treatment of youth anxiety:

1. Comparative Effectiveness: What is the comparative effectiveness of therapist-led (telehelath, hybrid or office-based) versus guided online formats of CBT to treat youth anxiety presenting to pediatric usual care settings?
2. Heterogeneity of Treatment Effects: Are there key factors that predict or moderate differential treatment engagement or response? Such factors, in turn, can inform treatment personalization for various patient subgroups, and ultimately more patient-centered care for pediatric anxiety.
3. What are the barriers and facilitators to delivering these treatment comparators in pediatric usual care settings and for the diverse patient populations served?

ELIGIBILITY:
To maximize generalizability, inclusion criteria were wider and exclusion criteria were minimal compared to majority of previous RCTs of youth anxiety treatment

Inclusion Criteria

1. Children age 7-18 years at the time of screening
2. Child has elevated anxiety as indicated by a T-score above 55 (greater than 0.5 SD (Standard Deviation) above the mean) on the PROMIS Item Bank v2.0 - Anxiety - Short Form 8a (child self-report or parent proxy report) in English or Spanish at the time of screening
3. Child and caregiver(s) are fluent in English or Spanish
4. Child's parent or legal guardian is age 16 or older
5. If child taking SSRI/Pharmacotherapy for anxiety, must be on stable dose for greater than or equal to 8 weeks from the time of screening (self-reported, must be reported by parent if under the age of 18)
6. Receiving care at sites participating in the study

Exclusion Criteria

1. Severity requiring higher level of care, as indicated by any of the following: (a) suicidal thoughts or behaviors (STP) with an active plan; (b) STB(s) requiring higher level of care in the past 6 months; (c) anxiety-related absence > 50% of school days over the past month (if summer, the last month of school enrolled); (d) substance use that required emergency services or inpatient/partial hospitalization within past 3 months; or (e) clinician-determination that child requires higher level of care.
2. History of diagnosed autism spectrum disorder with severe challenges and needs for support (e.g., complete absence of verbal communication unrelated to anxiety), or intellectual disability with severe challenges or needs for support.
3. Currently engaged in CBT or planning to continue a non-study psychotherapy for anxiety during the time of the study (self-reported, must be reported by parent if under the age of 18)
4. Treatment participants not fluent in English or Spanish
5. Child is ward of the state

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 305 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Comer, PhD, Principal Investigator — Florida International University; Donna B Pincus, PhD, Principal Investigator — Boston University
Locations (8):
- United States (8):
  - Nicklaus Children's Hospital, Miami, Florida
  - Florida International University, Miami, Florida
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - South Boston Community Health Center, Boston, Massachusetts
  - Harborview Medical Center, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Patient-Centered Outcomes Data Repository will be used to facilitate responsible sharing of principal data from the trial for appropriate secondary use.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will post by Dec 31, 2025. Will be available for at least 7 years (until Dec 30, 2032).
Access Criteria: Will be posted for public access and use on the Patient-Centered Outcomes Data Repository.
URL: https://www.icpsr.umich.edu/web/pages/pcodr/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment numbers refer to # of dyads, not # of individuals--that is, a treated child and their caregiver together count as 1 enrollment. Values in table below refer to # of dyads.
Period: Baseline
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Started | 156 | 149
Completed | 156 | 149
Not Completed | 0 | 0
Period: Midtreatment
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Started | 156 | 149
Completed | 112 | 123
Not Completed | 44 | 26
Not completed — Lost to Follow-up | 16 | 7
Not completed — Withdrawal by Subject | 28 | 19
Period: Posttreatment
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Started | 112 | 123
Completed | 112 | 118
Not Completed | 0 | 5
Not completed — Lost to Follow-up | 0 | 5
Period: Follow-up
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Started | 112 | 118
Completed | 80 | 94
Not Completed | 32 | 24
Not completed — Lost to Follow-up | 19 | 18
Not completed — Withdrawal by Subject | 13 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered) | Total
Number analyzed (Participants) | 156 | 149 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] — Child Age (continuous)
  years | 11.8 (2.8) | 12.0 (2.8) | 11.9 (2.8)
Age, Continuous [Mean (Standard Deviation); unit: years] — Caregiver Age (continuous)
  years | 42.65 (6.9) | 42.07 (6.5) | 42.37 (6.7)
Age, Customized [Count of Participants; unit: Participants] — Child Age Groups
  Participants
    7-12 years old | 104 | 99 | 203
    13-18 years old | 52 | 50 | 102
Sex/Gender, Customized [Count of Participants; unit: Participants] — Child Gender/Sex
  Participants
    Cis Male | 52 | 56 | 108
    Cis Female | 102 | 85 | 187
    Trans or NonBinary | 2 | 8 | 10
Sex/Gender, Customized [Count of Participants; unit: Participants] — Caregiver Sex/Gender
  Participants
    Female | 133 | 125 | 258
    Male | 13 | 13 | 26
    Not Reported | 10 | 11 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Child Race/Ethnicity. Note- Caregiver Race/Ethnicity data was not collected.
  Participants
    Hispanic/Latine | 71 | 70 | 141
    Hispanic/Latine & Asian | 3 | 1 | 4
    Hispanic/Latine & American Indian/Alaskan Native | 2 | 1 | 3
    Non-Hispanic White | 50 | 50 | 100
    Black or African American | 14 | 8 | 22
    Black & Hispanic/Latine | 4 | 5 | 9
    Black & American Indian/Alaskan Native | 0 | 1 | 1
    Black & Hispanic/Latine & American Indian/Alaskan Native | 0 | 1 | 1
    Black & Asian | 0 | 1 | 1
    Black & Middle Eastern/North African | 0 | 1 | 1
    Asian | 8 | 7 | 15
    Asian & Middle Eastern/North African | 0 | 1 | 1
    American Indian/Alaskan Native | 1 | 0 | 1
    American Indian/Alaskan Native & Native Hawaiian/Other Pacific Islander | 0 | 1 | 1
    Middle Eastern or North African (MENA) | 1 | 0 | 1
    Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 156 | 149 | 305
Caregiver Nativity [Count of Participants; unit: Participants]
  Caregiver U.S. Born | 92 | 93 | 185
  Caregiver Foreign Born | 64 | 56 | 120
Household Resource Insecurity [Count of Participants; unit: Participants] — Coded as having 'household resource insecurity' if the caregiver indicated that the family experienced any of the following over the past 12 months: (i) unhoused or living in a shelter, (ii) unable to pay the rent or mortgage on time, (iii) the food they purchased did not last and they did not have money to get more, (iv) there was concern their food would run out before they got money to buy more, and/or (v) the gas or electric company threatened to shut off or refuse gas or electricity to the house for not paying bills.
  Participants
    Baseline Household Resource Insecurity | 28 | 34 | 62
    No Baseline Household Resource Insecurity | 128 | 115 | 243
Non-English Language Spoken in Home [Count of Participants; unit: Participants]
  Yes | 82 | 79 | 161
  No | 73 | 68 | 141
  Not reported | 1 | 2 | 3
Caregiver Education [Count of Participants; unit: Participants]
  High School or Less | 58 | 61 | 119
  Completed College | 46 | 39 | 85
  Completed Graduate School | 41 | 37 | 78
  Not reported | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Promis Pediatric Short Form v. 2.0-Anxiety (Parent Proxy/Caregiver Report)
Description: This caregiver-report anxiety questionnaire is a publicly available measure that assesses youth fear, anxiety, misery, hyper-arousal, and somatic symptoms related to arousal. It also assesses behavioral fear avoidance. The form is available in English and Spanish and has excellent reliability and validity. The form includes 8 items and uses a scale of 1-5 (1=Never, 2=Almost never, 3= Sometimes, 4=Often, 5=Almost always). The raw score is the sum of the points for each response (range: 8-40), with higher scores represents higher levels of anxiety. Raw scores are converted to T-scores (range: 33.5-88.3), with higher T-scores representing higher levels of anxiety. T-scores of 50 reflect the population mean with a standard deviation of 10. Scores of 55 indicated elevated anxiety and >=60 reflecting clinical levels of anxiety. T scores are reported here and were subjected to analyses.
Time Frame: Baseline, Midtreatment (on average, 8 weeks), Posttreatment (on average, 19 weeks), Follow-up (on average, 55 weeks)
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 156 | 149
T-Score
  Baseline | 65.7 (8.3) | 66.0 (8.3)
  Midtreatment: number analyzed (Participants) | 112 | 123
  Midtreatment | 59.2 (9.4) | 59.1 (9.4)
  Posttreatment: number analyzed (Participants) | 112 | 118
  Posttreatment | 57.9 (9.7) | 57.7 (9.7)
  Follow-up: number analyzed (Participants) | 80 | 94
  Follow-up | 56.2 (10.2) | 55.9 (10.2)

2. Primary Outcome: Promis Pediatric Short Form v. 2.0-Anxiety (Pediatric/Youth Self-Report)
Description: This youth self-report anxiety questionnaire is a publicly available measure that assesses youth fear, anxiety, misery, hyper-arousal, and somatic symptoms related to arousal. It also assesses behavioral fear avoidance. The form is available in English and Spanish and has excellent reliability and validity. The form includes 8 items and uses a scale of 1-5 (1=Never, 2=Almost never, 3= Sometimes, 4=Often, 5=Almost always). The raw score is the sum of the points for each response (range: 8-40), with higher scores represents higher levels of anxiety. Raw scores are converted to T-scores (range: 33.5-88.3), with higher T-scores representing higher levels of anxiety. T-scores of 50 reflect the population mean with a standard deviation of 10. Scores of 55 indicated elevated anxiety and >=60 reflecting clinical levels of anxiety. T scores are reported here and were subjected to analyses.
Time Frame: Baseline, Midtreatment (on average, 8 weeks), Posttreatment (on average, 19 weeks), Follow-up (on average, 55 weeks)
Population: Intention-to-treat analyses
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 156 | 149
T scores
  Baseline | 61.4 (9.5) | 61.2 (9.5)
  Midtreatment: number analyzed (Participants) | 112 | 123
  Midtreatment | 55.6 (9.6) | 56.4 (9.6)
  Posttreatment: number analyzed (Participants) | 112 | 118
  Posttreatment | 54.7 (9.4) | 54.4 (9.4)
  Follow-up: number analyzed (Participants) | 80 | 94
  Follow-up | 54.4 (10.0) | 54.2 (10.0)

3. Primary Outcome: Child Anxiety Life Interference Scale (CALIS), Caregiver Report
Description: The Child Anxiety Life Interference Scale (CALIS) parent-report is a measure of caregiver perceptions of life interference and impairment associated with child anxiety. The CALIS has demonstrated strong psychometric properties, and assesses impairments in family, peer, academic, and extracurricular life domains. The CALIS parent-report 16 items administered to caregivers. All items, which relate to common activities (e.g. "being with friends outside of school" or "your career choice"), are rated on a five-point Likert scale (0 = not at all, 4 = a great deal), with higher scores indicating higher anxiety life interference. Scores range from 0-64.
Time Frame: Baseline, Midtreatment (on average, 8 weeks), Posttreatment (on average, 19 weeks), Follow-up (on average, 55 weeks)
Population: Intention-to-treat analyses
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 156 | 149
score on a scale
  Baseline | 26.3 (12.2) | 26.8 (12.2)
  Midtreatment: number analyzed (Participants) | 112 | 123
  Midtreatment | 20.2 (12.1) | 20.5 (12.1)
  Posttreatment: number analyzed (Participants) | 112 | 118
  Posttreatment | 18.9 (12.) | 19.3 (12.2)
  Follow-up: number analyzed (Participants) | 80 | 94
  Follow-up | 17.3 (12.2) | 17.6 (12.2)

4. Primary Outcome: Child Anxiety Life Interference Scale (CALIS), Youth Self-Report
Description: The Child Anxiety Life Interference Scale (CALIS) youth-report is a measure of youth self-reports of life interference and impairment associated with child anxiety. The CALIS has demonstrated strong psychometric properties, and assesses impairments in family, peer, academic, and extracurricular life domains. The CALIS youth self-report 9 items. All items, which relate to common activities (e.g. "being with friends outside of school" or "your career choice"), are rated on a five-point Likert scale (0 = not at all, 4 = a great deal), with higher scores indicating higher anxiety life interference. Scores range from 0-36.
Time Frame: Baseline, Midtreatment (on average, 8 weeks), Posttreatment (on average, 19 weeks), Follow-up (on average, 55 weeks)
Population: Intention-to-treat analyses
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 156 | 149
score on a scale
  Baseline | 13.1 (7.5) | 13.4 (7.5)
  Midtreatment: number analyzed (Participants) | 112 | 123
  Midtreatment | 10.6 (7.1) | 11.1 (7.1)
  Posttreatment: number analyzed (Participants) | 112 | 118
  Posttreatment | 10.6 (7.5) | 10.1 (7.5)
  Follow-up: number analyzed (Participants) | 80 | 94
  Follow-up | 9.5 (8.1) | 10.0 (8.1)

5. Secondary Outcome: Caregiver Treatment Satisfaction (Continuously Scored)
Description: To assess Caregivers Treatment Satisfaction, caregivers were administered a Satisfaction Scale that had them rate three items along 0-3 rating scales at at posttreatment: "Overall, how satisfied [have you been/were you] with the services that your family received?" [0=quite dissatisfied; 3=very satisfied]; "Would you recommend this program to a friend if they had a child with anxiety?" [0=no, definitely not; 3=yes, definitely]; and "How pleased [have you been/were you] with how this program has helped your child with anxiety" [0=quite displeased; 3=very pleased]. These three items were averaged for each informant to generate a Caregiver Total Satisfaction Score (range: 0-3, higher scores reflect greater satisfaction).
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat model means
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
score on a scale | 2.2 (0.7) | 2.7 (0.7)

6. Secondary Outcome: Caregiver Treatment Dissatisfaction (% of "Dissatisfied" Caregivers, Based on Dichotomous Coding of Dissatisfaction)
Description: At posttreatment caregivers were asked to rate three items developed for the present trial along 0-3 rating scales: "Overall, how satisfied were you with the services that your family received?" [0=quite dissatisfied; 3=very satisfied]; "Would you recommend this program to a friend if they had a child with anxiety?" [0=no, definitely not; 3=yes, definitely]; and "How pleased were you with how this program helped your child with anxiety" [0=quite displeased; 3=very pleased]. These items were averaged for each informant to generate a Caregiver Total Satisfaction Score (range: 0-3, higher scores reflect greater treatment satisfaction). For interpretation, mean scores <2 were interpreted as "Dissatisfied." Here we present the % of "Dissatisfied" caregivers at Post, across conditions.
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat
Measure: Number; unit: percentage of caregivers
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
percentage of caregivers | 23.9 | 6.8

7. Secondary Outcome: Youth Treatment Satisfaction (Continuously Scored)
Description: To assess Youth Treatment Satisfaction, youth > 8 years were administered a Satisfaction Scale that had them rate three items along 0-3 rating scales at posttreatment: "Overall, how satisfied [have you been/were you] with the services that you received?" [0=quite dissatisfied; 3=very satisfied]; "Would you recommend this program to a friend if they had anxiety?" [0=no, definitely not; 3=yes, definitely]; and "How pleased [have you been/were you] with how this program has helped you with anxiety" [0=quite displeased; 3=very pleased]. These three items were averaged for each informant to generate a Youth Total Satisfaction Score (range: 0-3, higher scores reflect greater satisfaction).
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat model means
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
score on a scale | 2.1 (.8) | 2.4 (.8)

8. Secondary Outcome: Youth Treatment Dissatisfaction (% of "Dissatisfied" Youth, Based on Dichotomous Coding of Dissatisfaction)
Description: At posttreatment, youth were asked to rate three items developed for the present trial along 0-3 rating scales: "Overall, how satisfied were you with the services that you received?" [0=quite dissatisfied; 3=very satisfied]; "Would you recommend this program to a friend if they had anxiety?" [0=no, definitely not; 3=yes, definitely]; and "How pleased were you with how this program helped your anxiety" [0=quite displeased; 3=very pleased]. These items were averaged for each informant to generate a Youth Total Satisfaction Score (range: 0-3, higher scores reflect greater treatment satisfaction). For interpretation, mean scores <2 were interpreted as "Dissatisfied." Here we present the % of "Dissatisfied" youth at Post, across conditions.
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat
Measure: Number; unit: percentage of youth
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
percentage of youth | 33.3 | 19.9

9. Secondary Outcome: Caregiver-Perceived Effectiveness
Description: To assess Caregiver-Perceived Effectiveness, caregivers were asked on a 7-point scale "How effective do you think the program [has been/was] in treating your child's anxiety?" [0=very ineffective; 3=somewhat effective; 6=very effective]. Range of possible scores: 0-42; higher scores reflect greater perceived effectiveness.
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat model means
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
score on a scale | 2.9 (1.8) | 4.2 (1.8)

10. Secondary Outcome: Rate of Treatment Responders (% of Children Whose Posttreatment PARS Score Was at Least 35% Less Than Their Baseline PARS Score)
Description: "Treatment Responder" defined as score reduction of at least 35% on the Pediatric Rating Scale (PARS). The PARS is a well-established clinician-rated instrument for assessing the frequency and severity of anxiety symptoms. Six global items are summed to generate a PARS Total score. The PARS has shown strong psychometric properties. PARS Total Score reductions of 35% or more are empirically defined as reflecting "Treatment Response". For the present study, PARS interviews were conducted by independent evaluators masked to treatment condition. Values here reflect the % of "Treatment Responders" at post, across conditions
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat
Measure: Number; unit: percentage of children
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
percentage of children | 48.7 | 55.4

11. Secondary Outcome: Caregiver Homework Engagement (% of Weeks Caregiver Completed Assigned Homework)
Description: Therapists completed weekly logs reporting whether study families on their caseloads completed the homework assigned in their previous session or support call. Homework completion reflects the percent of weeks across the trial in which all assigned homework was completed by caregiver, accounting for nesting and for covariates.
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat
Measure: Number; unit: percentage of trial weeks
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
percentage of trial weeks | 53.1 | 70.7

12. Secondary Outcome: Youth Homework Engagement (% of Weeks Youth Completed Assigned Homework)
Description: Therapists completed weekly logs reporting whether study families on their caseloads completed the homework assigned in their previous session or support call. Homework completion reflects the percent of weeks across the trial in which all assigned homework was completed by child/teen, accounting for nesting and for covariates.
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat
Measure: Number; unit: percentage of trial weeks
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
percentage of trial weeks | 50.8 | 61.9

13. Secondary Outcome: Treatment Completion (% of Children Who Completed Their Treatment Program)
Description: Therapists completed weekly logs reporting whether study families on their caseloads attended their scheduled sessions. Treatment Completion was defined for Therapist-Led CBT as attending 10 treatment sessions, and for Guided Online CBT Care as attending 4 support calls. For Guided Online CBT families, administrative backend data was also collected from the central server to further assess user/usage analytics. Values reflect % of completers within each condition.
Time Frame: Posttreatment (on average, 19 weeks)
Measure: Number; unit: percentage of children
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 156 | 149
percentage of children | 53.2 | 46.3

14. Secondary Outcome: Treatment Comprehension Difficulties (Caregiver Report)
Description: Caregivers were asked at Posttreatment "How hard has the intervention been for [your family/your child] and you to understand?" [0=never hard; 3=sometimes hard; 6=very hard]. This item was developed for the present study (range: 0-6), with higher scores reflecting greater comprehension difficulties.
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat model means
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
units on a scale | 1.67 (1.5) | 1.01 (1.1)

15. Secondary Outcome: Difficulty Making Time for Treatment (Caregiver Report)
Description: To assess Difficulties Making Time for Treatment caregivers were asked at at Posttreatment "How hard has it been for [your family/your child] to [make your schedule work for treatment sessions/find time to work on and complete the computer-based treatment modules online]?" [0=never a problem; 3=sometimes a problem; 6=often a problem]. This item was developed for the present study (range: 0-6), with higher scores reflecting greater difficulties making time for treatment.
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat model means
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
units on a scale | 3.17 (2.1) | 2.14 (1.8)

16. Secondary Outcome: Treatment Discomfort (Caregiver Report)
Description: Caregivers were asked at Posttreatment "How comfortable has your [family/child] felt when [attending treatment sessions/completing the computer-based treatment modules online]?" [0=very comfortable; 3=sometimes comfortable; 6=very uncomfortable]. This item was developed for the present study (range: 0-6), with higher scores reflecting greater treatment discomfort.
Time Frame: Posttreatment (on average, 19 weeks)
Population: Intention-to-Treat model means
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
Number analyzed (Participants) | 112 | 118
units on a scale | 2.81 (2.2) | 2.86 (2.6)

ADVERSE EVENTS:
Time Frame: 55 weeks
Description: Adverse Events in participating children were assessed, but Adverse Events were not assessed in participating caregivers.
Arm/Group | Guided Online CBT (With Minimal Therapist Involvement) | Therapist-Led CBT (Telehealth, Office-based, or Hybrid Delivered)
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/149
Other Adverse Events (participants affected / at risk) | 0/156 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT03707158/Prot_SAP_000.pdf